CLINICAL TRIAL: NCT00841724
Title: Phase II Study of a Reduced-toxicity " Submyeloablative " Conditioning Regimen Prior to Allogeneic Stem Cell Transplantation in Patients With Hematological Malignancies
Brief Title: Study of a Reduced-toxicity "Submyeloablative" Conditioning Regimen Prior to Allogeneic Stem Cell Transplantation in Patients With Hematological Malignancies
Acronym: ITT 08-01
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Anne Omnès, Nantes University Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRD 08/9-P
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Last update posted 2012-05-16 (Estimated); Status verified 2012-05

CONDITIONS: Hematological Malignancies
Keywords: Allogeneic stem cell transplantation; Reduced-intensity conditioning; Reduced-toxicity conditioning; Hematological malignancies; IV Busulfan
MeSH Terms: conditions — Hematologic Neoplasms | interventions — fludarabine; Busulfan; Antilymphocyte Serum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Busilvex, Fludara, Thymoglobuline (Active Comparator): D-6: Fludara D-5: Fludara + Busilvex D-4: Fludara + Busilvex D-3: Fludara + Busilvex D-2: Fludara + Thymoglobuline D-1: Thymoglobuline D0: graft infusion
  Interventions: Drug: Fludarabine, Busulfan, Thymoglobuline

INTERVENTIONS:
Drug: Fludarabine, Busulfan, Thymoglobuline

SUMMARY:
The goal of this prospective study is to assess the overall mortality (whether related to relapse/progression or toxicity - TRM-) at one year after allogeneic stem cell transplantation prepared by a so-called reduced-toxicity "submyeloablative" conditioning regimen in patients with hematological malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Patients affiliated to a social security reimbursement system
* Adults (men or women) aged between 18 and 65 years
* Negative test for pregnancy
* ECOG 0-1 or Karnofsky Index ≥ 70%
* Availability of an HLA-identical sibling donor, or an HLA-matched unrelated donor (10/10 HLA compatibility in A, B, C, DRB1, DQB1 (a single allelic mismatch at the level of Cw can be accepted)
* Life expectancy > 6 months
* Signed informed consent
* Diagnosis of an hematological malignancy that is considered to be eligible for an allogeneic stem cell transplantation

Exclusion Criteria:

* Pregnant woman or not willing to take effective contraception
* Classical contra-indications to the allogeneic stem cell transplantation procedure
* Any contra-indication to the use of the drugs contained within the conditioning regimen according to the summary of product characteristics
* Patients aged < 50 years and deemed to be eligible for a "standard" or conventional myeloablative conditioning regimen
* An HLA-matched sibling donor who has a contra-indication for stem cell mobilization and collection
* History of uncontrolled psychiatric condition
* Patients who have participated to another trial testing an experimental drug within one month prior to inclusion in this protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2009-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of the overall mortality rate at 12 months after allogeneic stem cell transplantation | 12 months after transplantation

SECONDARY OUTCOMES:
To assess the "classical" criteria (clinical and biological) associated with outcome after allogeneic stem cell transplantation. To evaluate the impact of the modified Charlson comorbidity score (Sorror Score) on TRM and 1-year overall survival | 12 months after transplantation

CONTACTS AND LOCATIONS:
Overall Officials: Mohamad Mohty, MD, PhD, Principal Investigator — Nantes University Hospital
Locations (3):
- France (3):
  - Institut Paoli Calmettes, Marseille
  - CHU de Nantes, Nantes
  - CHU de Bordeaux, Pessac